CLINICAL TRIAL: NCT04548453
Title: Establish the uSI Values and End-user Training Material That Will be Used to Guide Oxytocin Dosing Actions
Acronym: uSI-ranges
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: PreTeL, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: uSI range setting study
Record Dates: First submitted 2020-09-01; First posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Pregnancy Related; Labor Long; Fetal Distress
Keywords: labor; oxytocin; tachysystole; prolonged labor
MeSH Terms: conditions — Fetal Distress

STUDY DESIGN:
Intervention Model Description: prospective, non-significant risk
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Uterine EMG during labor (Experimental): Multichannel uterine electromyography will be recorded on patients receiving oxytocin for induction or augmenation of labor.
  Interventions: Device: uterine electromyography

INTERVENTIONS:
Device: uterine electromyography — Multichannel uterine electromyography will record uterine biosignals during labor.
  Other Names: electrohysterography

SUMMARY:
Patients receiving oxytocin for induction or augmentation of labor will be studied with uterine EMG. The results of the EMG will be converted to an oxytocin-associated uterine stimulation index (uSI), which is intended to guide decisions for changing the dose of oxytocin. An expert panel will review the results of the oxytocin dosing actions, then assigned optimized actions throughout the labor. The uSI will be correlated with the optimal dosing actions.

DETAILED DESCRIPTION:
Background. Oxytocin stimulates the uterus, increases the strength and frequency of uterine contractions and facilitates delivery. The "dose" of oxytocin is the rate of IV infusion. In a typical labor where oxytocin is used, many dosing adjustments are performed over many hours. Finding the correct dose for a given patient is challenging because some women respond rapidly to low doses of oxytocin, others require high doses. The correct dose is important because the risks of adverse outcomes increase when doses are either too low or excessive. The dosing actions increase, hold, decrease or stop are typically performed every 30 minutes during oxytocin administration.

Dosing actions are performed based on the current level of simulation caused by the current dose. To assess the level of stimulation, current methods rely heavily on the output of the fetal monitor, which produces contraction frequency and fetal heart rate. Additional information for dosing decisions is obtained from subjective assessments such uterine palpation. Subjective measures are used because there is no objective method available to reliably guide a dosing action. Subjectivity is a major contributor to the long duration of labor for inductions and the high rate of excessive uterine stimulation with any oxytocin use.

The uterine stimulation index (uSI) is an objective measure of the current level of stimulation caused by the current dose of oxytocin in individual patients and can be used to guide oxytocin dosing actions. uSI is based on an electromyography (EMG) signal that is proportional to the effects of oxytocin on the uterine muscle. uSI is calculated from multichannel EMG to obtain a representative sampling of the effects of oxytocin on entire uterus. The range of values for uSI is from 0 (no oxytocin effects) to 10 (maximal oxytocin effects). Low values of uSI guide the end-user to increase the current dose of oxytocin. Intermediate values of uSI guide the end-user to hold the current dose. High values of uSI guide the end-user to decrease the current dose.

The purpose of this study is to establish the ranges of uSI values that correspond to the dosing actions increase, hold and decrease. To establish these ranges, 51 subjects will undergo current methods of dosing while having multichannel EMG recorded. uSI values will not be available to end-users, so all subjects will receive dosing actions determined by standard of care using current method. After delivery, a panel of experts will retrospectively assess each dosing action based on the outcome of the dosing action. These "optimized dosing actions" will then be correlated with the uSI value obtained at that time. This process produces paired data of optimized actions and uSI values. From the clustering of the uSI values, the ranges of uSI can be matched to the dosing actions increase, hold and decrease.

As a second goal, human factors will be studied with questionnaires and end-user interviews to improve the methods used for recording multichannel EMG during labor.

Procedure. Patients receiving oxytocin for clinical indications will be approached for participation. After obtaining consent, up to 8 proprietary EMG sensors will be placed over the subject's abdomen, spanning most of the surface of the uterus. Additionally, one ground sensor and one noise rejection sensor will be placed. Multichannel EMG recordings will be obtained throughout the labor, although the results of the EMG will not be available to the obstetrical providers. Subjects will be managed using current methods of monitoring and standard of care for oxytocin dosing decisions.

At the conclusion of the recording, the EMG sensors will be removed from the subject. Data will be analyzed after delivery, producing uSI values as a function of time for the duration of the labor.

An expert panel will be assembled, composed of clinicians trained in the art of obstetrics and managing oxytocin. The progress of labor will be assessed by examining the fetal monitor strip (i.e. uterine contractile activity and the fetal heart rate over time), cervical changes, and the dosing actions performed. No less than 72 hours after delivery the neonate's and subject's medical records will be reviewed to identify complications of the delivery that may have occurred.

The expert panel will assess each dosing action as optimal or not optimal. An example of a not optimal action would be increasing the dose and causing uterine tachysytole. In this example, "hold" will be assigned as the optimized dosing action. Each subject will have a list of optimized dosing actions and the time they were performed. Optimized dosing actions will then be linked with uSI values observed at that time, creating a paired data set of uSI values and optimal dosing actions.

The optimized dosing actions increase, hold and decrease will be correlated with uSI values and the range of uSI values that correspond with each dosing action will be established.

End-users will be interviewed 1 to 72 hours after delivery of the baby. The interview will identify barriers to EMG recording may influence the effectiveness of the information provided by the multichannel EMG recording.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or greater
* At least 37 weeks gestation
* English reading and speaking
* Female gender
* Singleton fetus
* Planned continuous external fetal monitoring: to include fetal heart rate and uterine contraction monitoring
* May have clinical indications for internal monitoring (IUPC and/or FSE) that replaces external monitoring.
* Induction or augmentation of labor with oxytocin (Pitocin)
* Subjects undergoing artificial rupture of membranes (AROM) or who experienced spontaneous rupture of membranes (SROM), with a plan for oxytocin administration, will be included as a special category.
* Subjects may undergo cervical ripening.
* Patients must be able to review and sign informed consent to participate in the study.
* Trial of labor after Cesarean section are eligible for participation
* Women diagnosed with diabetes and/or pre-eclampsia with or without magnesium therapy are eligible for participation
* Women with other complications of pregnancy are eligible for participation if the complication does not interfere with fetal monitoring, EMG monitoring or other recording of data.

Exclusion Criteria:

* Non-English reading and/or speaking
* Twins, triplets and other multifetal gestations
* Non-vertex presentation
* Planned Cesarean delivery
* Significant uterine anomalies such as didelphys or bicornuate uterus (women with small, clinically insignificant anomalies such as uterine fibroids are not excluded).
* Participants cannot be participating in any other research study or protocol regarding uterine contraction monitoring during the same study period as required for our study.
* Known allergy to ECG pad adhesive
* Non-living fetus
* Major fetal malformation
* Fetal distress, or other indications for emergent delivery
* Other than a Category I fetal heart tracing at the beginning of the recording.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All subjects will be pregnant, hence will be women
Enrollment: 51 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Correlating uSI with the optimized dosing actions increase, hold and decrease | 8 months
  uSI clustering with dosing actions will be identified to provide guidance when prospectively dosing oxytocin
Human factors in recording multichannel EMG during labor | 8 months
  Difficulties and discomfort of the EMG recording process will be identified and corrected

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers. Data in summary form, based on numerical assessments of the uSI and optimized dosing actions will be published.